CLINICAL TRIAL: NCT06622031
Title: Transjugular Intrahepatic Portosystemic Shunt Combined With Lenvatinib and PD-1 Inhibitor for Advanced Hepatocellular Carcinoma With Main Trunk Portal Vein Tumor Thrombus: a Multicenter Phase II Study
Brief Title: TIPS Combined With Lenvatinib and PD-1 Inhibitor for Advanced HCC With Main Trunk PVTT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qunfang, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liver Projiect 11
Record Dates: First submitted 2024-09-30; First posted 2024-10-01 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus; Systemic Therapy
Keywords: Advanced hepatocellular carcinoma; Lenvatinib; Sintilimab; Camrelizumab; Tislelizumab; Transjugular intrahepatic portosystemic shunt; Main trunk portal vein tumor thrombus
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Portasystemic Shunt, Transjugular Intrahepatic; lenvatinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Intervention Model Description: TIPS procedure
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transjugular intrahepatic portosystemic shunt (Experimental): A needle punctured the portal vein through the transjugular approach. After a successful puncture, the parenchymal tract was dilated, and covered stents were introduced. The specifications of the covered stents were 8 mm × 50 mm, 8 mm × 60 mm, 8 mm × 70 mm, and 8 mm × 80 mm. All of the diameters of the bare stents were 8 mm, and the lengths were 50-80 mm. The portal vein pressure was measured before and after shunt creation. After the insertion of TIPS, all of the participants received a diuretic treatment and a salt-limited diet.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt; Drug: Lenvatinib; Drug: PD-1 inhibitor

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt — A needle punctured the portal vein through the transjugular approach. After a successful puncture, the parenchymal tract was dilated, and covered stents were introduced. The specifications of the covered stents were 8 mm × 50 mm, 8 mm × 60 mm, 8 mm × 70 mm, and 8 mm × 80 mm. All of the diameters of the bare stents were 8 mm, and the lengths were 50-80 mm. The portal vein pressure was measured before and after shunt creation. After the insertion of TIPS, all of the participants received a diuretic treatment and a salt-limited diet.
  Other Names: TIPS
Drug: Lenvatinib — 12 mg (body weight ≥60 kg) , 8 mg (body weight <60 kg
Drug: PD-1 inhibitor — Tislelizumab (200mg intravenously every 3 weeks), Sintilimab (200mg intravenously every 3 weeks), Camrelizumab (200mg intravenously every 3 weeks)

SUMMARY:
Hepatocellular carcinoma (HCC) with main trunk portal vein tumor thrombus (PVTT) has poor prognosis. The main lethiferous factor is the upper gastrointestinal hemorrhage by PVTT-related portal hypertension, then the second is the tumor-caused death. It is vital to prevent the portal hypertension by PVTT.

DETAILED DESCRIPTION:
Portal hypertension by main trunk portal vein tumor thrombus (PVTT) is a severe disease. Patients usually die of gastrointestinal hemorrhage rather than tumor progression. It is vital to prevent the portal hypertension. Transjugular intrahepatic portosystemic shunt (TIPS) is an effective method to alleviate the portal pressure. Then the risk of gastrointestinal hemorrhage is decreased which provides an opportunity for system therapy. In this study, the investigators explore the TIPS combined with Lenvatinib and PD-1 inhibitor for advanced hepatocellular carcinoma with main trunk portal vein tumor thrombus. The investigators aim to add clinical evidence for this subtype of advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of primary HCC, confirmed histologically or clinically according to the criteria of the American Association for the Study of Liver Diseases;
2. presence of PVTT with III-IV grade by Cheng's criteria;
3. having PVTT induced portal hypertension;
4. with or without PVTT induced acute variceal bleeding;
5. metastases with limited five sites and no more two organs involved;
6. Number of Intrahepatic tumors were no more than five;
7. receipt of Lenvatinib and PD-1 inhibitor as the first-line systemic therapy;
8. classified as Child-Pugh class A or B and having an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 2;
9. no history of other malignancies;
10. agreed to participated in this clinical trial;
11. Hemameba ≥3.0 x109/L, neutrophil ≥1.5x109/L, hemoglobin≥10.0 g/L, platelet≥100x 109/L, ALT; AST; bilirubin ≤1.5-fold normal, GFR≥60ml/min.

Exclusion Criteria:

1. recurrent HCC;
2. PVTT at I-II grade by Cheng's criteria;
3. age < 18 years or > 75 years;
4. advanced HCC with more than five metastases;
5. Number of Intrahepatic tumors were more than five;
6. no response to Lenvatinib;
7. life expectancy less than 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Rates of gastrointestinal hemorrhage | 6 months
  atients occur gastrointestinal hemorrhage within 6 months after TIPS.

SECONDARY OUTCOMES:
Progression-Free-Survival (PFS) | 12 months
  Progression was defined as progressive disease by independent radiologic review
Overall survival (OS) | 24 months
  OS is the length of time from the date of inclusion until death from any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all included patients whose best overall response (BOR) is either a complete response or partial response.
Adverse events | 24 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations

CONTACTS AND LOCATIONS:
Overall Officials: Feng Duan, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General hospital, Beijing, None Selected, China